CLINICAL TRIAL: NCT05385237
Title: Noninvasive Stage Identification of Hepatic Fibrosis Using 4D-MRI
Brief Title: Identification of Hepatic Fibrosis Using 4D-MRI
Acronym: 4D-MRI Liver
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2020-02669; th22Bieri
Record Dates: First submitted 2022-05-17; First posted 2022-05-23 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Liver Diseases
Keywords: Magnetic resonance imaging (MRI); non-alcoholic fatty liver (NAFLD); alcohol-related liver disease (ALD); elastography; liver deformation; liver stiffness; liver fibrosis
MeSH Terms: conditions — Liver Diseases; Non-alcoholic Fatty Liver Disease; Liver Cirrhosis

STUDY DESIGN:
Intervention Model Description: prospective, national, multi-center study
Who Masked: Outcomes Assessor
Masking Description: Statistician blinded for analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4D-MRI assessment for patients with liver diseases (Experimental): patients with chronic liver diseases, acute liver inflammation or cardiac blood congestion to the liver will be assessed by MRI
  Interventions: Diagnostic Test: 4D-MRI
- 4D-MRI assessment for healthy volunteers (control group) (Experimental): healthy control subjects will be assessed by MRI
  Interventions: Diagnostic Test: 4D-MRI

INTERVENTIONS:
Diagnostic Test: 4D-MRI — Novel MR-imaging (MRI) and postprocessing techniques, making it possible to capture breathing-induced abdominal motion, including liver motion, under free-breathing. For the first time, these techniques - called 4D-MRI - were able to capture the abdominal organs with high spatial resolution in 3-dimensions at a high frame rate of 2-3 Hz and enabled an entirely new insight into the human body.

SUMMARY:
To date, no specific treatment options exist for liver diseases, and there is a large global effort to find drugs that will halt liver disease progression in these patients.Liver fibrosis staging is essential as a diagnostic/prognostic measure and there is an increasing demand for accurate non-invasive liver stiffness measurement tools. This research project proposes a novel MR-based quantitative Liver Deformation Biomarker (qLDB) approach for non-invasive liver fibrosis assessment by using a new technique called 4D-MRI. 4D-MRI allows to overcome the limitations of currently used techniques. Hence, 4D-MRI may help to identify a novel biomarker for non-invasive staging of liver fibrosis , and therefore improve the final diagnosis of patients suffering from liver diseases.

DETAILED DESCRIPTION:
Chronic liver diseases represent a rising global health threat. A prolonged inflammatory state leads to progressive fibrosis that can result in liver cirrhosis associated with serious complications including loss of liver function or hepatocellular carcinoma development. A particularly strong increase in the prevalence, morbidity, and mortality occurs in fatty liver disease, such as non-alcoholic fatty liver disease (NAFLD) and alcohol-related liver disease; (ALD).To date, no specific treatment options for these conditions exist, and there is a large global effort to find drugs that will halt liver disease progression in these patients. Liver fibrosis staging is essential as a diagnostic/prognostic measure and there is an increasing demand for accurate non-invasive liver stiffness measurement tools. This research project proposes a novel MR-based quantitative Liver Deformation Biomarker (qLDB) approach for non-invasive liver fibrosis assessment by using a new technique called 4D-MRI. This technique makes it possible to overcome limitations in currently used techniques, i.e. to capture the abdominal organs with high spatial resolution in 3-dimensions at a high frame rate of 2-3 Hz and enabled an entirely new insight into the human body. The final diagnosis (i.e., stage of fibrosis) is based on quantifying changes of the liver's mechanical properties by dynamic magnetic resonance (MR) measurements and comparing the liver's elastic deformation with healthy livers. This innovative methodology allows for the first time to quantitatively measure the elastic deformation of organs during free-breathing and for an extended period, since no harmful X-rays are required. The hypothesis of the study is that the mechanical changes a liver undergoes during liver disease progression are visible in 4D-MRI data sets as a reduced elasticity. This will be assessed using our 4D-MRI approach taking into account the liver's deformation induced by natural respiration and also cardiac pulsation. The primary objective of the study is to compare liver deformation, induced at different respiratory breath-hold positions, by respiratory motion, and cardiac pulsation, between healthy subjects and patients with histologically confirmed liver cirrhosis in order to find a novel biomarker for non-invasive staging of liver fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* (a) Patients with histologically confirmed chronic liver disease, including NAFLD, ALD, viral hepatitis B and C, genetic (e.g. Wilson disease, hemochromatosis) or autoimmune liver disease
* (b) Patients with acute liver inflammation or cardiac blood congestion to the liver (as assessed by laboratory values, imaging findings and clinical history)
* ability to understand and consent to participate in this study

Exclusion Criteria:

* Medical implant like cardiac pacemaker, pump, hip prosthesis
* Metallic objects in the body (e.g. splinters after an accident)
* Persons who have undergone brain or cardiac surgery
* Claustrophobia
* Body Weight >140kg or as provided by the MR manufacturer
* Pregnant and lactating women
* (a) Active hepatocellular carcinoma (HCC) (remark: patients with a history of HCC and curative treatment can be included)
* (a) CHILD C cirrhosis
* (a) and (b) Patients with overt ascites (except if they respond to diuretic treatment and the ascites resolves)
* (c) Metabolic syndrome, BMI >30 kg/m2
* (c) Acute or chronic liver disease
* Patients not willing or able to give a written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the spatial-temporal deformation fields | 90 days
  To find out whether the spatial-temporal deformation fields, as induced by natural respiration and cardiac pulsation, and as assessed by dynamic MR measurements, are changed in liver cirrhosis if compared to healthy livers.

SECONDARY OUTCOMES:
Assessment of mechanical changes with 4D-MRI | 90 days
  To assess whether the mechanical changes a liver undergoes during liver disease progression are visible in 4D-MRI data sets as a progressively reduced elasticity, and can be correlated to histological data of the study participants
Differential Diagnosis | 90 days
  To assess whether the liver's mechanical properties/elastic deformation can differentiate between liver fibrosis (due to chronic liver disease) and acute inflammatory processes/venous blood congestion
Superiority Assessment of 4D-MRI vs.US elastography | 90 days
  To assess whether 4D-MRI shows improved sensitivity and specificity if compared to US-elastography in staging hepatic fibrosis
Superiority Assessment of 4D-MRI vs, standard MRI | 90 days
  To assess whether 4D-MRI shows improved sensitivity and specificity if compared to standard clinical liver MRI in staging hepatic fibrosis

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Filipowicz Sinnreich, PD Dr., Principal Investigator — University Hospital of Basel
Locations (2):
- Switzerland (2):
  - Kantonsspital Baselland (KSL), Liestal, Basel-Landschaft
  - University Hospital Basel, Basel, Canton of Basel-City

IPD SHARING:
Plan to Share IPD: Undecided